CLINICAL TRIAL: NCT00878761
Title: Randomized Double-Blind, Placebo-Controlled, Single and Multiple Dose, Dose-Escalation Study of STX 100 in Renal Transplant Patients With Biopsy Proven Interstitial Fibrosis and Tubular Atrophy (IF/TA)
Brief Title: Study of STX-100 in Renal Transplant Patients With Interstitial Fibrosis and Tubular Atrophy (IF/TA)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Stromedix, Inc. (Industry)
Responsible Party: Bradley Maroni, MD, Stromedix, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STX-002
Record Dates: First submitted 2009-04-06; First posted 2009-04-09 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Chronic Allograft Dysfunction
Keywords: Renal transplant; Interstitial fibrosis and tubular atrophy; Chronic allograft dysfunction; Chronic allograft nephropathy; kidney transplant
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- STX-100 (0.03mg/kg) (Experimental): 8 patients (6 active and 2 placebo)
  Interventions: Biological: STX-100
- STX-100 (0.1mg/kg) (Experimental): 8 patients (6 active and 2 placebo)
  Interventions: Biological: STX-100
- STX-100 (0.3mg/kg) (Experimental): 16 patients (12 active and 4 placebo)
  Interventions: Biological: STX-100
- STX-100 (1mg/kg) (Experimental): 16 patients (12 active and 4 placebo)
  Interventions: Biological: STX-100

INTERVENTIONS:
Biological: STX-100 — SC, single dose followed by multiple dose

SUMMARY:
This Phase 2 study is a multi-center, randomized, double-blind, placebo-controlled, single followed by multiple dose, dose escalation study designed to evaluate the safety, tolerability, pharmacokinetics, immunogenicity, and impact of STX-100 on gene and protein expression for αvβ6 related and TGF-β-inducible genes (including tubulointerstitial injury, epithelial function, and IF/TA related genes) in renal transplant patients with biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adult patients, 18 (or the legal age of consent) to 65 years old, male or female.
* eGFR ≥ 25 ml/min (Cockcroft-Gault formula).
* Six to 60 months post renal transplant at the initiation of screening.
* Qualifying renal biopsy obtained within 8 weeks prior to randomization with histologic evidence of ≥ Grade 2 IF/TA (Banff score) without morphologic evidence of a treatable etiology (e.g., BK virus nephropathy, chronic obstruction).
* Adequate bone marrow and liver function
* Weight between 40-110 kg.
* Female patients must be surgically sterile, postmenopausal (minimum 1 year without menses and verified by follicular-stimulating hormone [FSH] levels), or agree to use contraception from the time of signing the informed consent form through 16 weeks following the last injection of study medication. Male patients must also agree to use birth control for either themselves or their partner, as appropriate, from the time of signing the informed consent form through 16 weeks following the last injection of study medication.

Exclusion Criteria:

* Recipient of a multi-organ transplant.
* History of T-cell mediated rejection (TCMR) within 3 months prior to randomization.
* Patients who are receiving high dose corticosteroids at the time of screening.
* Histologic evidence of acute TCMR (≥ Banff Grade 1A) on a qualifying renal biopsy for this study. Patients with 'borderline' changes (Banff criteria) on a qualifying renal biopsy are eligible for this study if the Principal Investigator believes treatment for TCMR is not warranted.
* Prior or current histologic evidence of polyomavirus BK virus nephropathy.
* Any histologic finding on the qualifying renal biopsy that the Investigator believes warrants modifying the patient's current therapy.
* Evidence of active tissue invasive cytomegalovirus or Epstein-Barr virus infection.
* History of malignancy, including carcinoma or post-transplant lymphoproliferative disorder.
* History of chronic pulmonary disease or smoker within the past 5 years or more than 15 pack-years exposure.
* Serious local infection or systemic infection within 3 months prior to screening.
* Surgery within 3 months prior to Day 1 (other than minor cosmetic surgery, minor dental procedures, or percutaneous kidney transplant biopsy).
* Positive test for HBsAg, HCV, or HIV antibody at screening.
* Treatment with another investigational drug, investigational device, or approved therapy for investigational use within 1 month prior to dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by adverse events | 25 weeks from first dosing (per cohort)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Maroni, MD, Study Chair — Stromedix, Inc.
Locations (1):
- Stromedix Investigative Site, Cambridge, Massachusetts, United States